CLINICAL TRIAL: NCT05921708
Title: Examination of Physical Activity, Exercise Preferences, Body Image, and Social Media Usage Behaviors of X, Y, and Z Generation Women
Brief Title: The Examination of Woman Generations' on Exercise Preferences, Body Image, Physical Activity and Social Media Use
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Rabia Sanir, Lecturer PT, Istanbul University - Cerrahpasa
Other Study IDs: 2023/38
Record Dates: First submitted 2023-06-18; First posted 2023-06-27 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Healthy Woman; Body Image
Keywords: physical activity; social media; exercise; physical appereance; generational difference
MeSH Terms: conditions — Motor Activity | interventions — Telemedicine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- X Generation: Generation X refers to those born between 1965 and 1979 (1).
  Interventions: Other: Assessment1; Other: Assesment2; Other: Assessment3; Other: Assessment4; Other: Assessment5
- Y Generation: Generation Y is a population, also known as the Millennials, who was born between 1980 and 1994 (1).
  Interventions: Other: Assessment1; Other: Assesment2; Other: Assessment3; Other: Assessment4; Other: Assessment5
- Z Generation: Generation Z are individuals born between 1995 and 2015 (1).
  Interventions: Other: Assessment1; Other: Assesment2; Other: Assessment3; Other: Assessment4; Other: Assessment5

INTERVENTIONS:
Other: Assessment1 — International Physical Activity Questionnaire (IPAQ) (Short)
  Other Names: International Physical Activity Questionnaire (IPAQ) (Short)
Other: Assesment2 — Physical Appearance Comparison Scale-Revised (PACS-R)
  Other Names: Physical Appearance Comparison Scale-Revised (PACS-R)
Other: Assessment3 — Sociocultural Attitudes Towards Appearance Questionnaire -4-Revised (SATAQ-4R)
  Other Names: Sociocultural Attitudes Towards Appearance Questionnaire -4-Revised (SATAQ-4R)
Other: Assessment4 — Body-Cathexis Scale (BCS)
  Other Names: Body-Cathexis Scale (BCS)
Other: Assessment5 — Mobile Health, Exercise Preferences and Social Media Questionnaire
  Other Names: Mobile Health, Exercise Preferances and Social Media Questionnaire

SUMMARY:
Purpose: The aim of this study is to examine the differences in the physical activity levels, exercise preferences, body image, and social media use of the women of the X, Y, and Z generations and to determine the relationship between these parameters and the use of social media.

Method Type of study: This research is a descriptive cross-sectional study and the population of the study consists of women. Evaluations of the participants will be made in the form of an online survey via "Google Forms".

Participants: The sample size of the study was calculated using the G Power program with the One Way Anova method, with a type 1 error value of α=0.05, power (1-ß)= 0.90, and effect size (predicted)=0.25 to be at least 207 individuals. The women constituting the sample of the study will be divided into three different groups X-Y-Z according to the generations based on the stratified random sampling method.

DETAILED DESCRIPTION:
Intervention: The groups will be compared in terms of their physical activity levels, exercise preferences, body image, body image, and their relationship with social media use will be examined. In this study, the International Physical Activity Questionnaire (IPAQ) (Short), Physical Appearance Comparison Scale-Revised (PACS-R), Sociocultural Attitudes Towards Appearance Questionnaire -4-Revised (SATAQ-4R), Body-Cathexis Scale (BCS) and Mobile health scale created by researchers in line with the purpose of the research. and Social Media Usage and Exercise Preferences questionnaire will be used.

Statistical Analysis: SPSS (Statistics Program for Social Sciences) 26.0 will be used for statistical analysis. The suitability of the data to the normal distribution will be evaluated with the Kolmogorov-Smirnov test. Descriptive statistics will be shown as mean ± standard deviation, minimum and maximum value for continuous variables, and categorical variables will be shown as frequency and percentage. Chi-square analysis will be used to compare categorical variables. The data of the 3 groups will be compared statistically. If the data has a normal distribution, parametric tests will be preferred, and if the data is not normally distributed, nonparametric tests will be preferred. In all statistical analyses, p<0.05 or 95% confidence interval will be accepted as the level of significance.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years or older
* Female gender
* Birth year range to be between 1965 and 2005
* Being a volunteer for attending the study

Exclusion Criteria:

* Having any musculoskeletal injury within 6 months
* Having any neurological, rheumatological, or cardiac problems
* Having a psychiatric illness

Ages: 18 Years to 58 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Generation X refers to those born between 1965 and 1979 Generation Y, also known as the Millennials, born between 1980 and 1994 Generation Z are individuals born between 1995 and 2015
Sampling Method: Probability Sample
Enrollment: 230 (Estimated)
Dates: Start 2023-06-30 (Estimated); Primary Completion 2023-07-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Sociocultural Attitudes Towards Appearance Questionnaire -4-Revised (SATAQ-4R) | 1 month, June 2023- July2023
  The SATAQ-4R created by Schaefer, Harriger et al., consists of 31 items and seven sub-parameters: body fat, muscle level, general attractiveness, peers, family, others, and media (2).
Physical Appearance Comparison Scale-Revised (PACS-R) | 1 month, June 2023- July2023
  It was developed to measure a person's tendencies to compare their physical appearance with the physical appearance of others. The survey consists of 11 questions. It includes questions that assess whether it compares body shape, body weight, and body fat in social settings, such as at the gym, at work, or at school (3).

SECONDARY OUTCOMES:
Mobile Health, Exercise Preferances and Social Media Questionnaire | 1 month, June 2023- July2023
  The attitudes of the participants towards mobile health applications and their social media usage habits will be evaluated with the Mobile Health and Social Media Usage questionnaire created by the researchers. The survey will question the frequency of use of social media, purposes of use, platforms, the mobile application used, frequency of use and purposes of use. Participants' attitudes towards their exercise preferences will be evaluated with the Exercise Preferences questionnaire, and their regular exercise habits, preferred exercise type, environment and method will be questioned.
International Physical Activity Questionnaire (IPAQ) (Short) | 1 month, June 2023- July2023
  International Physical Activity Questionnaire (IPAQ) (Short) is a 7-item scale that evaluates the duration and frequency of vigorous physical activity, moderate physical activity, walking and sedentary behavior based on MET values (4).
Body-Cathexis Scale (BCS) | 1 month, June 2023- July2023
  The scale consists of 40 items, each of which is related to an organ or a part of the body or its function. Items are scored between 1-5. While the most positive statement receives one point and the most negative statement receives five points, the lowest total score that can be obtained from the scale, which has an answer option such as "I like it very much", "I like it very much", "I am undecided", "I don't like it very much", "I don't like it at all", is 40, and the highest is 40. The total score is 200. An increase in the total score obtained from the scale means an increase in negative evaluation, while a decrease in the score indicates positive evaluation (5).

CONTACTS AND LOCATIONS:
Overall Officials: Rabia SANIR, Study Chair — Istanbul University Cerrahpasa- Halic University; Ayşenur NAMLI SEKER, Study Chair — Istanbul University - Cerrahpasa; Ipek YELDAN KARAGOZ, Study Director — Istanbul University - Cerrahpasa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Betz CL. Generations X, Y, and Z. J Pediatr Nurs. 2019 Jan-Feb;44:A7-A8. doi: 10.1016/j.pedn.2018.12.013. No abstract available. PMID 30683288
- [Background] Schaefer LM, Harriger JA, Heinberg LJ, Soderberg T, Kevin Thompson J. Development and validation of the sociocultural attitudes towards appearance questionnaire-4-revised (SATAQ-4R). Int J Eat Disord. 2017 Feb;50(2):104-117. doi: 10.1002/eat.22590. Epub 2016 Aug 19. PMID 27539814
- [Background] Schaefer LM, Thompson JK. The development and validation of the Physical Appearance Comparison Scale-Revised (PACS-R). Eat Behav. 2014 Apr;15(2):209-17. doi: 10.1016/j.eatbeh.2014.01.001. Epub 2014 Feb 4. PMID 24854806
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Kundakçı, A. H. (2005). Comparison of University Students in terms of Eating Attitudes, Self Perceptions, Body Image and Stress Symptoms, Master Thesis, Ankara University Institute of Social Sciences, Ankara.